CLINICAL TRIAL: NCT01271738
Title: Measuring the Effect of Additional Tumor Cavity Margins Excision at the Time of Breast Conserving Surgery for Stage 0, I, II, and III Breast Cancer Patients on Re-excision Rate, Cosmetic Results and Total Costs
Brief Title: Evaluating and Comparing Two Surgical Methods for Treatment of Early Stage Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Monica Rizzo, Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00013658; WCI1659-09 (Other: Other)
Record Dates: First submitted 2010-12-06; First posted 2011-01-07 (Estimated); Last update posted 2015-08-17 (Estimated); Status verified 2015-08

CONDITIONS: Breast Neoplasms; Breast Cancer; Breast Tumors; Cancer of Breast; Cancer of the Breast; Human Mammary Carcinoma; Neoplasms, Breast
Keywords: Breast Cancer; Tumors or cancer of the human breast; Breast Tumors; Cancer of Breast; Cancer of the Breast; Human Mammary Carcinoma; Neoplasms, Breast
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — Histocompatibility Testing

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Breast Conserving Surgery (BCS) (Active Comparator)
  Interventions: Procedure: Remove tumor only
- Breast Conserving Surgery with Additional 5 Margins (BCS + M) (Active Comparator)
  Interventions: Procedure: Removal of tumor and tissue

INTERVENTIONS:
Procedure: Remove tumor only — No additional margins (tissue) removed at the initial surgery
  Arms: Breast Conserving Surgery (BCS)
Procedure: Removal of tumor and tissue — 5 additional margins (tissue) removed at the time of surgery
  Arms: Breast Conserving Surgery with Additional 5 Margins (BCS + M)

SUMMARY:
The goal of this study is to compare two different types of breast surgery. In the first type, the doctor removes only the tumor. In the second type, the doctor removes the tumor and some of the tissue around the tumor called margins. The amount of breast tissue removed is similar. The removal of the tumor only has up to 40% chance of reoperation because the tumor is too close to the margin. The primary goal of this study is to see if the additional margins can decrease the need to return to the operating room. Both types of surgery are well accepted, and participating in the study would not give you a better chance to cure the cancer. At present, most breast surgeons remove the tumor without the additional margins. For all patients who have this operation, there is a high incidence of return to the operating room for margins re-excision: as many as 40% as patients can have a re-operation.

At present, we do not know if taking the additional margins prevents the cancer from returning in the breast or not. If the cancer comes back in your breast, this is a recurrence and your breast will have to be removed (mastectomy).

ELIGIBILITY:
Inclusion Criteria:

* Female Patients with the diagnosis of Stage 0, I, II and III breast cancer diagnosed/treated at the AVON Foundation Comprehensive Breast Center (AFCBC) of Grady Memorial Hospital
* Age: no limit

Exclusion Criteria:

* Stage IV breast cancers

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2009-09; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Comparing 2 surgical methods for treatment of early stage breast cancer | Post operative evaluation will be at 30 days, then at 4-7 months and last at 12-15 months.
  The investigator will survey patients with the cosmetic assessment survey after the surgical procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Monica Rizzo, MD, Principal Investigator — EmoryUniversity Winship Cancer Institute
Locations (1):
- Emory University Winship Cancer Institute, Atlanta, Georgia, United States